CLINICAL TRIAL: NCT06461676
Title: Study of Intramyocardial Injection of Ventrix Bio Extracellular Matrix (VentriGel) to Assess the Safety and Feasibility in Pediatric Patients with Hypoplastic Left Heart Syndrome (HLHS)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Ventrix, Inc. (Industry); University of California, San Diego (Other)
Responsible Party: Principal Investigator, William T. Mahle, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006965
Record Dates: First submitted 2024-05-28; First posted 2024-06-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Stage II Glenn operation; HLHS
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ventrix Bio Extracellular Matrix (Experimental): Treatment intervention of a total of 8 injections into the right ventricle of the heart will occur before the patient comes off of the heart-lung bypass machine used during the Stage II Glenn Operation. The treatment will be conducted according to clinical guidelines set in place while the patient is undergoing a surgical intervention before the patient comes off the heart/lung bypass machine required for the stage II Glenn Procedure.
  Interventions: Drug: Ventrix Bio Extracellular Matrix

INTERVENTIONS:
Drug: Ventrix Bio Extracellular Matrix — VentriGel will be administered by injection into the right ventricle of the heart in the following defined doses per injection. There will be a total of 8 injections. The proposed dose of up to 0.6 mL is administered as up to 8 sequential injections of 4 injections of 0.1 mL each and 4 injections of 0.05 mL each.
  Other Names: VentriGel

SUMMARY:
The goal of this Phase I Open-Label study is to demonstrate the safety and feasibility of VentriGel injection in children with Hypoplastic Left Heart Syndrome (HLHS).

The main questions it aims to answer are:

* Whether VentriGel is safe in treating patients with HLHS
* Whether there are any preliminary improvements in measures of cardiac function following Ventrigel injection

DETAILED DESCRIPTION:
HLHS, a type of congenital heart disease, presents a unique challenge where the left ventricle fails to develop, necessitating the right ventricle to manage both systemic and pulmonary blood flow. This condition, once fatal, has become manageable due to advancements in surgical techniques, with reported 5-year survival rates of 70-90%. However, these staged procedures, while lifesaving, can strain the right ventricle, leading to long-term issues such as weakened muscle and reduced cardiac function. Additionally, even with surgical intervention, patients often face a diminished quality of life.

Addressing these challenges, ongoing clinical trials explore regenerative therapies, particularly stem cell injections, aiming to improve heart function. Yet, concerns persist regarding the practicality and efficacy of these treatments, including issues with cell survival and coordination of injections within narrow timeframes.

Innovatively, the investigator and the team propose an alternative approach using VentriGel, an injectable hydrogel derived from decellularized porcine myocardium. Originally designed for treating heart failure post-myocardial infarction in adults, VentriGel has shown promising results in animal models, demonstrating significant improvements in cardiac function. Notably, its shelf-stable nature and flexible timing for administration offer advantages over traditional stem cell therapies.

Moreover, VentriGel's effectiveness in addressing right-ventricular failure, as demonstrated in recent studies, highlights its potential as a solution for HLHS patients. Leveraging approved extracellular matrix devices, such as Alloderm and SurgiSIS, further underscores the feasibility and safety of this approach, paving the way for potentially transformative treatments in congenital heart diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Hypoplastic Left Heart Syndrome (HLHS) requiring Stage II Glenn operation under one year of age

Exclusion Criteria:

* Subjects undergoing the Stage II Glenn operations who do not have HLHS
* Subjects requiring mechanical circulatory support within 5 days pre pre-surgical intervention
* Parent or guardian unwilling or unable to comply with necessary follow-up(s)
* Immunosuppressive diseases or subjects who require treatment with interventions that cause immunosuppression
* A history of tumor or malignancy
* Coagulation disorders
* Chromosomal abnormalities that limit expected survival to < 1 year
* Abnormal lab values that may increase the risk of the study procedure (WBC >20,000 cells/ul or < 1,000 cells/ul; platelet count < 50,000 cells/ul; Hgb < 8.0 gm/dl; LFTs > 2x reference lab upper limit of normal) at the time of screening
* Subjects with conduction abnormalities, including atrioventricular block and bundle branch blocks
* Ventricular arrhythmias due to antiarrhythmic pharmacological therapy

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of ventricular tachycardia events | upto 30 days post operation
  Number of sustained/symptomatic ventricular tachycardia incidences requiring intervention with inotropic support or anti-arrhythmics
Number of Cardiogenic shock events | Day 1, 30 days post operation
  Cardiogenic shock (i.e. tissue hypoperfusion presented by hypotension due to decreased cardiac output, determined by rising lactate levels (5x normal levels in first 24 hours, 2.5x normal levels in first 30 days)
Number of unplanned cardiovascular operation events | 30 days post operation
  Unplanned cardiovascular operation due to right ventricular intramyocardial injection site bleeding in the first 5 days after Stage II operation decreased cardiac output, determined by rising lactate levels (5x normal levels in first 24 hours, 2.5x normal levels in first 30 days)
Number of patients requiring new permanent pacemaker | upto 30 days post operation
  Number of patients requiring new permanent pacemaker
Stroke or embolic event | upto 30 days post operation
  Stroke or embolic event to the brain determined by CT scan
Number of Adverse Events | upto 30 days post operation
  Number of adverse events occurring post op
Number of deaths | upto 30 days post operation
  Number of deaths occurring post op
Number of VentriGel products manufactured and delivered to subjects | 12 months
Number of patients receiving Cardiac MRIs | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Change in right ventricular ejection fraction | Baseline, 6 months, 12 months post operation
  This will be measured by serial echocardiograms and MRI scans
Change in right ventricular end diastolic volume | Baseline, 6 months, 12 months post operation
  This will be measured by serial echocardiograms and MRI scans
Change in right ventricular end systolic volume | Baseline, 6 months, 12 months post operation
  This will be measured by serial echocardiograms and MRI scans
Change in tricuspid regurgitation | Baseline, 6 months,12 months post operation
  This will be measured by serial echocardiograms and MRI scans. tricuspid regurgitation measured by tricuspid valve vena contracta width
Change in right ventricular function Fractional Area Change | Baseline, 6 months,12 months post operation
  This will be measured by serial transthoracic echocardiogram (TTE)
Change in right ventricular global longitudinal strain | Baseline, 6 months,12 months post operation
  This will be measured by serial transthoracic echocardiogram (TTE)
Change in right ventricular global circumferential strain | Baseline, 6 months,12 months post operation
  This will be measured by serial transthoracic echocardiogram (TTE)
Change in right ventricular Tricuspid Annular Plane Systolic Excursion (TAPSE) | Baseline, 6 months,12 months post operation
  This will be measured by serial transthoracic echocardiogram (TTE)
Change in right atrial volume indexed | Baseline, 6 months,12 months post operation
  This will be measured by serial transthoracic echocardiogram (TTE)

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Altanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No